CLINICAL TRIAL: NCT02260089
Title: A Multicenter Open-label Study of the Efficacy and Safety of Telmisartan in Mild to Moderate Hypertensive Patients
Brief Title: Telmisartan in Mild to Moderate Hypertensive Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 502.363
Record Dates: First submitted 2014-10-08; First posted 2014-10-09 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan

ARMS (2):
- Low dose of telmisartan (Experimental): 4 week placebo run-in phase followed by 6 weeks of treatment with low dose of telmisartan
  Interventions: Drug: Low dose of telmisartan; Drug: Placebo
- High dose of telmisartan (Experimental): After 6 weeks of treatment with low dose of telmisartan, titration to high dose of telmisartan if blood pressure level is higher than 140/90 mm Hg
  Interventions: Drug: High dose of telmisartan

INTERVENTIONS:
Drug: Low dose of telmisartan
  Arms: Low dose of telmisartan
Drug: High dose of telmisartan
  Arms: High dose of telmisartan
Drug: Placebo
  Arms: Low dose of telmisartan

SUMMARY:
To evaluate the efficacy and tolerability of telmisartan, given once a day to patients with mild to moderate hypertension, as well as to assess the 24-hour blood pressure profile with ABPM

ELIGIBILITY:
Inclusion Criteria:

* Patients with blood pressure levels of 140/90 mm Hg or higher (confirmed on 2 consecutive visits), who were 18 years old and older, regardless of sex

Exclusion Criteria:

* Suspected or known diagnosis of arterial hypertension with a secondary cause
* Women who were not using an effective method of contraception, or who were pregnant, or breast-feeding
* Systolic blood pressure > 200 mm Hg or diastolic blood pressure > 115 mm Hg
* Laboratory test values two fold above the upper normal limit
* Previous intolerance to angiotensin conversion enzyme inhibitors or angiotensin II blocker (AIIAR)
* New York Heart Association class III or IV heart failure
* History of stroke in the 6 months prior to entry into the study
* Uncontrolled type 2 diabetes mellitus, defined as fasting glucose levels > 140 mg/dL on 3 consecutive assessments
* Patients who were included in another investigational drug study in the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2000-03; Primary Completion 2002-07 (Actual)

PRIMARY OUTCOMES:
Changes in systolic blood pressure (SBP) and diastolic blood pressure (DBP) | Baseline, up to 12 weeks after start of treatment
  Blood pressure values were obtained 24 hours after the last dose (through values) at the office

SECONDARY OUTCOMES:
Assessment of treatment response for SBP/DBP (in %) | Baseline, up to 12 weeks after start of treatment
  Response categories:
  * SBP < 140 mm Hg or
  * DBP < 90 mm Hg or
  * BP reduction ≥ 10 mm Hg
Changes from baseline in blood pressure values | Baseline, up to 12 weeks after start of treatment
  Analysis performed for the ambulatory blood pressure monitoring (ABPM) - subgroup
Number of patients with adverse events | Up to 16 weeks
Number of patients with clinically significant changes in laboratory values | Up to 16 weeks
Number of patients with clinically significant changes in ECG | Up to 16 weeks